CLINICAL TRIAL: NCT02839148
Title: Assessment of Maternal Perception Regarding Childhood Stunting and Development of a Tool to Assess Appetite in Children
Brief Title: Development of Appetite Measuring Tool and Appetite Status of Stunted Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR-16005
Record Dates: First submitted 2016-06-29; First posted 2016-07-20 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2018-08

CONDITIONS: Nutritional Stunting
Keywords: Appetite, Stunting, Satiety, Children
MeSH Terms: conditions — Growth Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary supplementation (Experimental): In case of dietary supplementation, we will provide milk and egg 6 days a week for 3 months to stunted children.
  Interventions: Dietary Supplement: Food supplementation
- psychosocial stimulation (Experimental): In case of psychosocial stimulation, we well provide PS weekly for first month, fortnightly for 2nd and 3rd months and then monthly for next 3 months. The total number of visits will be 11 over a period of 6 months.
  Interventions: Dietary Supplement: Food supplementation

INTERVENTIONS:
Dietary Supplement: Food supplementation — Arm 1 will be given food supplementation (FS), psychosocial stimulation (PS) and routine clinical care will be given and arm will be provided only with routine clinical care.
  The control children will receive routine clinical care but no FS or PS.
  Other Names: Routine clinical care, psychosocial stimulation

SUMMARY:
This study will provide a tool for researchers to measure important outcomes in relation to trial of intervention to reduce or prevent stunting.

Hypothesis: We assume that appetite score will be associated with improvement in growth and development parameters of children given the nutrition and psychosocial stimulation intervention

Objectives:

To explore maternal perception regarding childhood stunting To develop and validate an appetite measuring tool To assess the appetite status of young children To examine the relationship between appetite score, growth and development, potential biomarkers of appetite, child food intake and intestinal inflammation of the children.

Methods: In the first phase, a qualitative study will be conducted to explore maternal perception regarding childhood stunting and to develop a tool- the "Early Childhood Appetite and Satiety Tool"(ECAST) using mixed method approach (qualitative and quantitative). In the second phase, a community-based trial will be conducted with 50 stunted children of aged 12-18 months, living in urban slums of Dhaka, and 50 age-sex matched control children (non-stunted).

DETAILED DESCRIPTION:
The stunted children will receive an intervention package which includes food supplementation (FS) with one egg and 150 ml of whole milk supplementing the usual home diet, 6 days a week for 3 months; psychosocial stimulation (PS) for 6 months, and routine clinical care monthly for 6 months. The control children will receive routine clinical care but no FS and PS. Routine clinical care includes micronutrients powder, de-worming, health and nutrition education and immunization. All children will be assessed for appetite score (ECAST score) and anthropometry-at baseline then monthly for 6 months; food intake at baseline then monthly for 3 months, and cognitive development using Bayley Scales of Infant and Toddler Development, third version (Bayley-III) on enrolment and at 3 and 6 months of enrolment. Blood samples will be collected to examine gut hormones, complete blood count and haemoglobin percentage.

Stool samples will be collected for routine examination and stool biomarkers. Urine sample will be collected for screening urinary tract infection. All the specimens will be collected at baseline and at 3 and 6 months of enrollment.

Outcome measures/variables:

The primary outcome:

Assessment of appetite score of stunted children aged 12-18 months compared to non-stunted children.

The secondary outcomes are:

-Association of appetite score with growth and development with potential biomarkers of appetite with child food intake and intestinal inflammation of the children.

ELIGIBILITY:
Inclusion Criteria:

* 50 stunted children (LAZ<-2) aged 12-18 months
* 50 non-stunted (LAZ≥-2) aged 12-18 months

Exclusion Criteria:

* Severe acute malnutrition (SAM)
* Chronic illness
* Congenital anomaly/developmental delay/oromotor dysfunction

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 390 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Assessment of appetite score of stunted children aged 12-18 months compared to non-stunted children | 4 months

SECONDARY OUTCOMES:
Association of appetite score with growth and development child food intake | 15 months
Association of appetite score with growth and potential biomarkers of appetite | 15 months
Association of appetite score with growth and intestinal inflammation of the children | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Baitun Nahar, PhD, Principal Investigator — Associate Scientist
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
if required we will share data with our expertise

REFERENCES:
- [Derived] Naila NN, Mahfuz M, Hossain M, Arndt M, Walson JL, Nahar B, Ahmed T. Improvement in appetite among stunted children receiving nutritional intervention in Bangladesh: results from a community-based study. Eur J Clin Nutr. 2021 Sep;75(9):1359-1367. doi: 10.1038/s41430-020-00843-9. Epub 2021 May 27. PMID 34045689
- [Derived] Hossain M, Nahar B, Haque MA, Mondal D, Mahfuz M, Naila NN, Gazi MA, Hasan MM, Haque NMS, Haque R, Arndt MB, Walson JL, Ahmed T. Serum Adipokines, Growth Factors, and Cytokines Are Independently Associated with Stunting in Bangladeshi Children. Nutrients. 2019 Aug 7;11(8):1827. doi: 10.3390/nu11081827. PMID 31394828